CLINICAL TRIAL: NCT02020278
Title: A Phase 3b, Multicenter, Extension Follow-up Trial to Evaluate the Long-term Safety of Children and Adolescent Subjects With Euvolemic or Hypervolemic Hyponatremia Who Have Previously Participated in a Trial of Titrated Oral SAMSCA® (Tolvaptan)
Brief Title: An Extension Follow-up Trial to Evaluate the Long-term Safety of Children and Adolescent Participants With Euvolemic or Hypervolemic Hyponatremia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Issues with recruitment and enrollment made the trial impossible or highly impracticable. Termination of this trial was not due to safety reasons.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-11-294
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Euvolemic; Hypervolemic; Serum sodium; Dilutional hyponatremia; Electrolyte abnormality; Electrolyte imbalance; Metabolic disease; Water-Electrolyte Imbalance
MeSH Terms: conditions — Hyponatremia; Metabolic Diseases; Water-Electrolyte Imbalance | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tolvaptan (Experimental): Participants enrolled in this trial were eligible to receive open-label tolvaptan if they had a clinical need as determined by the investigator and met the eligibility criteria for optional tolvaptan treatment.
  Daily dose levels would have included 3.75 milligrams (mg), 7.5 mg, 15 mg, 30 mg, and 60 mg.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan 3.75-, 7.5-, 15-, and 30-mg spray-dried tablets. Dosage: Depending on age and weight, Tablet (3.75 mg - 60 mg daily). Frequency: Once daily.
  Duration: Participants may be eligible to receive short-term or long-term optional tolvaptan treatment at any time during their participation in the trial, with one or more treatment cycles over a 6-month period.
  Other Names: SAMSCA®

SUMMARY:
The objective of this trial was to provide 6 months of safety follow-up for children and adolescents with dilutional (euvolemic or hypervolemic) hyponatremia who had previously participated in a tolvaptan hyponatremia trial and to assess the efficacy of tolvaptan in increasing serum sodium for those participants who received optional continuing tolvaptan treatment of variable duration (up to 6 months).

DETAILED DESCRIPTION:
Core Safety Follow-up Component

• For all participants: To evaluate the post-treatment safety follow-up of children and adolescent participants with dilutional (euvolemic or hypervolemic) hyponatremia who have previously participated in a tolvaptan hyponatremia trial.

Optional Tolvaptan Treatment Component

• For participants who receive optional tolvaptan treatment: To demonstrate that tolvaptan safely and effectively achieves and maintains increased serum sodium concentrations in children and adolescent participants with dilutional (euvolemic or hypervolemic) hyponatremia when used for both multiple short-term treatments, and/or longer chronic treatments.

ELIGIBILITY:
Core Safety Follow-up Component

Inclusion Criteria: Participation in a prior pediatric trial with tolvaptan for euvolemic or hypervolemic hyponatremia.

Exclusion Criteria: None

Optional Tolvaptan Treatment Component (per treatment cycle)

Eligibility Criteria:

1. Male and female participants ≥ 4 years of age (or per local Health Authority age restrictions) and ≥ 10 kilograms (kg).
2. Participant must have been off treatment with the investigational medicinal product for at least 7 days following the end of treatment in the previous tolvaptan trial for hyponatremia (euvolemic or hypervolemic).
3. Persistent dilutional (euvolemic or hypervolemic) hyponatremia defined as being documented as present for at least 48 hours, evidenced by at least 2 serum sodium assessments < 130 milliequivalents (mEq)/liter (L) (millimole [mmol]/L) drawn at least 12 hours apart (these values can be documented using historical values previously obtained per standard of care); a third (STAT) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for efficacy endpoints, had to be obtained within 2 to 4 hours prior to the first dose of tolvaptan.
4. Ability to swallow tablets.
5. Ability to maintain adequate fluid intake whether orally or via intravenous support with adequate monitoring.
6. Ability to comply with all requirements of the trial.
7. Trial-specific written informed consent/assent obtained from a parent/legal guardian or legally acceptable representative, as applicable per age of participant or local laws, prior to the initiation of any protocol-required procedures. In addition, the participant as required by local laws must provide informed assent at the pretreatment baseline for this trial and must be able to understand that he or she can withdraw from the trial at any time. All informed consent/assent procedures must be in accordance with the trial center's Institutional Review Board/Independent Ethics Committee and local regulatory requirements.
8. Ability to commit to remain fully abstinent (periodic abstinence [for example, calendar, ovulation, symptothermal, post-ovulation methods] or withdrawal are not acceptable methods of contraception) or practice double-barrier birth control during the trial and for 30 days following the last dose of IMP for sexually active females of childbearing potential.

Ineligibility Criteria:

1. Had evidence of hypovolemia or intravascular volume depletion (for example, hypotension, clinical evidence of volume depletion, response to saline challenge); if the participant had systolic blood pressure or heart rate outside of the normal range for that age, then volume status was to be specifically clinically assessed to rule out volume depletion.
2. Had serum sodium < 120 mEq/L (mmol/L), with or without associated neurologic impairment (that is, symptoms such as apathy, confusion, or seizures).
3. Use of potent CYP3A4 inhibitors in participants ≤ 50 kg or moderate CYP3A4 inhibitors in participants < 20 kg.
4. Lacked free access to water (inability to respond to thirst) or without ICU-level fluid monitoring and management.
5. Had a history or current diagnosis of nephrotic syndrome.
6. Had transient hyponatremia likely to resolve (for example, head trauma or post-operative state).
7. Had hyperkalemia defined as serum potassium above the upper limit of normal (ULN) for the appropriate pediatric age range.
8. Had estimated glomerular filtration rate (eGFR) < 30 milliliters (mL)/minute (min)/1.73 meters squared (m^2) calculated by the following equation: eGFR (mL/min/1.73 m^2) = 0.413 x height (centimeter [cm])/serum creatinine (mg/deciliter [dL]).
9. Had acute kidney injury defined as: Increase in serum creatinine by ≥ 0.3 mg/dL (≥ 26.5 micromoles [μmol]/L) within 48 hours; or increase in serum creatinine to ≥ 1.5 times baseline, which was known or presumed to have occurred within the prior 7 days; or urine volume < 0.5 mL/kg/hour for 6 hours.
10. Had severe or acute neurological symptoms requiring other intervention (for example, hyperemesis, obtundation, seizures).
11. Had had treatment for hyponatremia with:

    * Hypertonic saline (including normal saline challenge) within 8 hours of qualifying sodium assessments;
    * Urea, lithium, demeclocycline, conivaptan, or tolvaptan within 4 days of qualifying serum sodium assessments;
    * Other treatment for the purpose of increasing serum sodium concurrent with dosing of trial medication
12. Had anuria or urinary outflow obstruction, unless the participant was, or could be, catheterized during the trial.
13. Had a history of drug or medication abuse within 3 months prior to the pretreatment visit or current alcohol abuse.
14. Had a history of hypersensitivity and/or idiosyncratic reaction to benzazepine or benzazepine derivatives (such as benazepril).
15. Had psychogenic polydipsia (participants with other psychiatric illness may be included per medical monitor approval).
16. Had uncontrolled diabetes mellitus, defined as fasting glucose > 300 mg/dL (16.7 mEq/L [mmol/L]).
17. Had screening liver function values > 3 x ULN.
18. Had cirrhosis and met any of the following conditions: a major gastrointestinal bleed within the past 6 months, evidence of active bleeding (for example, epistaxis, petechiae/purpura, hematuria, or hematochezia), platelet count < 50,000/μL, or use of concomitant medications known to increase bleeding risk.
19. Had hyponatremia due to the result of any medication that can safely be withdrawn (for example, thiazide diuretics).
20. Had hyponatremia (for example, hyponatremia in the setting of adrenal insufficiency, untreated hypothyroidism, or hypotonic fluid administration) that is most appropriately corrected by alternative therapies.
21. Was currently pregnant or breastfeeding.
22. Had any medical condition that, in the opinion of the investigator, could interfere with evaluation of the trial objectives or safety of the participants.
23. Was deemed unsuitable for trial participation in the opinion of the investigator.
24. Participation in another investigational drug trial within the past 30 days, without prior approval from the sponsor medical monitor.
25. Participants < 4 years of age (or per local Health Authority age restrictions), weight < 10 kg, or who were unable to swallow tablets.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (11):
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Grand Rapids, Michigan
  - Kansas City, Missouri
  - New York, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Seattle, Washington
- Ghent, Belgium
- Prague, Czechia
- Germany (2):
  - Erlangen, Nurnberg
  - Leipzig, Saxony
- Italy (4):
  - Genova
  - Naples
  - Palermo
  - Rome
- Romania (2):
  - Bucharest
  - Sibiu
- Madrid, Spain
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Small studies with less than 25 participants are excluded from data sharing.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants included those enrolled in a previous tolvaptan pediatric trial for hyponatremia (NCT02012959); who provided written informed consent at baseline and were able to understand that he/she could withdraw at any time; with the ability to comply with all requirements of the trial; ready to be followed up for 6 months.
Pre-assignment Details: There was no screening phase. Approximately 100 male or female participants were planned to be enrolled in this trial. A total of 3 participants were enrolled in this trial, but no participant received optional investigational medicinal product during this trial.
Groups:
- Tolvaptan: All participants enrolled first entered a 6-month follow-up trial that evaluated post-treatment safety after participation in a tolvaptan hyponatremia trial. Participants were then eligible to receive open-label tolvaptan if they had a clinical need as determined by the investigator and met the eligibility criteria for optional tolvaptan treatment during the 6-month follow-up period. In this trial, no participants qualified for treatment during the 6-month follow-up period. Daily dose levels would have included 3.75 milligrams (mg), 7.5 mg, 15 mg, 30 mg, and 60 mg.
Period: Core Safety Follow-up Component
Arm/Group | Tolvaptan
Started | 3
Completed | 3
Not Completed | 0
Period: Optional Tolvaptan Treatment Component
Arm/Group | Tolvaptan
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants: No enrolled participant received any investigational medicinal product during the study. Due to the low number of participants enrolled, 0 participants are reported due to the risk of reidentification.
Groups:
- Tolvaptan: All participants enrolled first entered a 6-month follow-up trial that evaluated post-treatment safety after participation in a tolvaptan hyponatremia trial. Participants were then eligible to receive open-label tolvaptan if they had a clinical need as determined by the investigator and met the eligibility criteria for optional tolvaptan treatment during the 6-month follow-up period. In this trial, no participants qualified for treatment during the 6-month follow-up period. Daily dose levels would have included 3.75 mg, 7.5 mg, 15 mg, 30 mg, and 60 mg.
Arm/Group | Tolvaptan
Number analyzed (Participants) | 0
Age, Continuous [unit: years] — Population: Due to the low number of participants enrolled, 0 participants are reported due to the risk of re-identification.
Sex: Female, Male [unit: participants] — Population: Due to the low number of participants enrolled, 0 participants are reported due to the risk of re-identification.
Ethnicity (NIH/OMB) [unit: Participants] — Population: Due to the low number of participants enrolled, 0 participants are reported due to the risk of re-identification.
Race (NIH/OMB) [unit: Participants] — Population: Due to the low number of participants enrolled, 0 participants are reported due to the risk of re-identification.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline At Month 6 In Serum Sodium While Tolvaptan Was Being Administered
Description: No enrolled participant received any investigational medicinal product during the study. Due to early study termination, efficacy data were not collected for this outcome measure.
Time Frame: Baseline, Month 6
Population: No enrolled participant received any investigational medicinal product during the study. Due to early study termination, efficacy data were not collected.
Groups:
- Optional Tolvaptan Treatment Component: The duration for the optional tolvaptan treatment (referred to as optional tolvaptan treatment component) was to be case-specific. It could have been short-term or long-term and could have consisted of 1 or more treatment cycles. Eligibility for optional tolvaptan treatment was to be determined at the pretreatment baseline visit of each dosing cycle. Each tolvaptan treatment cycle was to include a titration phase of up to 4 days and interruption of tolvaptan for up to 2 doses after 30 (±1) days of tolvaptan treatment. Due to early study termination, no participant entered the Optional Tolvaptan Treatment Component of this study.
Arm/Group | Optional Tolvaptan Treatment Component
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage Of Participants Who Required Rescue Therapy While On Tolvaptan Treatment
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 1
Groups:
- Optional Tolvaptan Treatment Component: The duration for the optional tolvaptan treatment (referred to as optional tolvaptan treatment component) was case-specific. It could have been short-term or long-term and could have consisted of 1 or more treatment cycles. Eligibility for optional tolvaptan treatment was to be determined at the pretreatment baseline visit of each dosing cycle. Each tolvaptan treatment cycle was to include a titration phase of up to 4 days and interruption of tolvaptan for up to 2 doses after 30 (±1) days of tolvaptan treatment.
Arm/Group | Optional Tolvaptan Treatment Component
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage Of Participants Who Had Recurrence Of Hyponatremia While On Tolvaptan
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | Optional Tolvaptan Treatment Component
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage Of Participants Requiring Continuation Of Tolvaptan Following 30 Days Of Treatment
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | Optional Tolvaptan Treatment Component
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline In Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale (GCS) Total Score At Month 6
Description: The PedsQL GCS was used for quality of life assessment. It is appropriate for at least 2 years of age, however availability may be limited for certain ages and languages. It encompasses 4 dimensions of functioning (physical, emotional, social, school). The age groups covered are: Toddler (2-4 years), Young child (5-7 years), Child (8-12 years), and Adolescent (13-18 years). Depending on the participant's age, the questionnaire may be completed by either the participant or the parent/caregiver, as appropriate. For the Toddler group, the PedsQL GCS consists of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL GCS consists of 23 items, with a 3-point Likert scale (0, 2, 4) for the Young Child, and a 5-point Likert scale for the Child and Adolescent groups. Scores are transformed on a scale from 0 to 100 and averaged. Higher scores indicate improved quality of life. The change from baseline in the GCS total score is presented.
Time Frame: Baseline, Month 6
Population: All enrolled participants with analyzable data at specified timepoint. No enrolled participant received any investigational medicinal product during the study.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Core Safety Follow-up Component: The core safety follow-up component of the trial was a 6-month period in which pediatric participants (children and adolescents) with dilutional (euvolemic or hypervolemic) hyponatremia, who previously participated in a tolvaptan hyponatremia trial, were to be followed (at a clinical trial site and/or through telephone calls), regardless of the need for treatment for hyponatremia, to assess the long-term safety of tolvaptan.
Arm/Group | Core Safety Follow-up Component
Number analyzed (Participants) | 1
units on a scale | -3.5 [-3.5 to -3.5]

6. Secondary Outcome: Change From Baseline In PedsQL GCS Physical Health Summary Score At Month 6
Description: The PedsQL GCS was used for quality of life assessment. It is appropriate for at least 2 years of age, however availability may be limited for certain ages and languages. It encompasses 4 dimensions of functioning (physical, emotional, social, school). The age groups covered are: Toddler (2-4 years), Young child (5-7 years), Child (8-12 years), and Adolescent (13-18 years). Depending on the participant's age, the questionnaire may be completed by either the participant or the parent/caregiver, as appropriate. For the Toddler group, the PedsQL GCS consists of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL GCS consists of 23 items, with a 3-point Likert scale (0, 2, 4) for the Young Child, and a 5-point Likert scale for the Child and Adolescent groups. Scores are transformed on a scale from 0 to 100 and averaged. Higher scores indicate improved quality of life. The change from baseline in the physical health dimension is presented.
Time Frame: Baseline, Month 6
Population: as for outcome 5
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Core Safety Follow-up Component
Number analyzed (Participants) | 1
units on a scale | 12.5 [12.5 to 12.5]

7. Secondary Outcome: Change From Baseline In PedsQL GCS Psychosocial Health Summary Score At Month 6
Description: The PedsQL GCS was used for quality of life assessment. It is appropriate for at least 2 years of age, however availability may be limited for certain ages and languages. It encompasses 4 dimensions of functioning (physical, emotional, social, school). The age groups covered are: Toddler (2-4 years), Young child (5-7 years), Child (8-12 years), and Adolescent (13-18 years). Depending on the participant's age, the questionnaire may be completed by either the participant or the parent/caregiver, as appropriate. For the Toddler group, the PedsQL GCS consists of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL GCS consists of 23 items, with a 3-point Likert scale (0, 2, 4) for the Young Child, and a 5-point Likert scale for the Child and Adolescent groups. Scores are transformed on a scale from 0 to 100 and averaged. Higher scores indicate improved quality of life. The change from baseline in summed emotional, social, and school dimensions is presented.
Time Frame: Baseline, Month 6
Population: as for outcome 5
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Core Safety Follow-up Component
Number analyzed (Participants) | 1
units on a scale | -13.5 [-13.5 to -13.5]

8. Secondary Outcome: Change From Baseline In PedsQL Multidimensional Fatigue Scale (MFS) Total Score At Month 6
Description: as for outcome 7
Time Frame: Baseline, Month 6
Population: as for outcome 5
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Core Safety Follow-up Component
Number analyzed (Participants) | 1
units on a scale | 9.7 [9.7 to 9.7]

9. Secondary Outcome: Percentage Of Participants With Overly Rapid Correction In Serum Sodium 24 Hours After The First Dose At Introduction Or Reintroduction Of Tolvaptan
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 1
Arm/Group | Optional Tolvaptan Treatment Component
Number analyzed (Participants) | 0

10. Secondary Outcome: Plasma Concentrations Of Tolvaptan And Metabolites In Participants Who Had Continued Tolvaptan Therapy For Eight Consecutive Weeks
Description: as for outcome 1
Time Frame: 8 Weeks
Population: No enrolled participant received any investigational medicinal product during the study. Due to early study termination, no pharmacokinetic analyses were performed.
Arm/Group | Optional Tolvaptan Treatment Component
Number analyzed (Participants) | 0

11. Secondary Outcome: Participants With A Tanner Staging Score Of 1 At Month 6
Description: Tanner Staging assessment consists of 2 domains (pubic hair and breast development) for girls and 3 domains (pubic hair, penis development, and testes development) for boys. Staging was based on a single score summarizing the domains (not individual domain scores). Stages range from 1-5, with 1 indicating preadolescent and 5 adult. Participants with a Tanner staging score of 1 (preadolescent) at Month 6 are reported.
Time Frame: Month 6
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Core Safety Follow-up Component
Number analyzed (Participants) | 3
Participants | 2

12. Secondary Outcome: Change From Baseline In Growth Percentiles For Body Height And Weight At Month 6
Description: Changes from baseline in growth percentiles for body height and weight were calculated and are reported.
Time Frame: Baseline, Month 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Core Safety Follow-up Component
Number analyzed (Participants) | 3
percentile
  Height Percentile | 19.0 (40.0)
  Weight Percentile | 0.7 (8.0)

13. Secondary Outcome: Change From Baseline In Alanine Aminotransferase (ALT) And Aspartate Aminotransferase (AST) For Participants On Tolvaptan At Month 2
Description: No enrolled participant received any investigational medicinal product during the study. Due to early study termination, efficacy data were not collected. Data reported only include assessments made for ALT and AST during the Core Safety Follow-up Component of the trial. Results are reported in units/liter (U/L).
Time Frame: Baseline, Month 2
Population: All enrolled participants with analyzable data at specified timepoint. No enrolled participant received any investigational medicinal product during the study. Due to early study termination, efficacy data were not collected.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Core Safety Follow-up Component
Number analyzed (Participants) | 2
U/L
  ALT | -10.00 (45.25)
  AST | -7.50 (0.71)

14. Secondary Outcome: Change From Baseline In Bilirubin For Participants On Tolvaptan At Month 2
Description: No enrolled participant received any investigational medicinal product during the study. Due to early study termination, efficacy data were not collected. Data reported only include assessments made for bilirubin during the Core Safety Follow-up Component of the trial. Results are reported in micromoles (umol)/L.
Time Frame: Baseline, Month 2
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Core Safety Follow-up Component
Number analyzed (Participants) | 2
umol/L | 2.57 (3.63)

ADVERSE EVENTS:
Time Frame: Baseline to Month 6
Arm/Group | Tolvaptan
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=3)
Pyrexia (General disorders) | 1
Enterovirus Infection (Infections and infestations) | 1
Rhinovirus Infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (N=3)
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Enterovirus Infection (Infections and infestations) | 1
Rhinovirus Infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
This trial was prematurely terminated due to challenges in enrollment. The trial was not terminated due to safety reasons. Due to early termination of the study, no efficacy data were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2015-11-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT02020278/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02020278/SAP_001.pdf